CLINICAL TRIAL: NCT05959135
Title: Ultrasound Evaluation of Gastric Content in Diabetic and Non-Diabetic Term Pregnant Women: An Observational Study
Brief Title: Gastric Ultrasound in Diabetic and Non-Diabetic Pregnant Women
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, KAIRATBEK MIIZAMOV, Principal Investigator, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 709654
Record Dates: First submitted 2023-07-07; First posted 2023-07-25 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Gastric Ultrasonography; Gastric Volume; Pulmonary Aspiration; Diabetic Pregnancy; Fasting
Keywords: Diabetic Pregnant Women; Gastric ultrasonography; Gastric Contents; Gastric volume; Antral sectional area; Pregnant women
MeSH Terms: conditions — Diabetes, Gestational; Fasting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic term pregnant patients: Compare the antral cross-sectional area (CSA) with gastric ultrasonography and estimated gastric volumes calculated with Perlas and Roukhomovsky mathematical models
  Interventions: Device: Gastric ultrasonography
- Non-Diabetic term pregnant patients: Compare the antral cross-sectional area (CSA) with gastric ultrasonography and estimated gastric volumes calculated with Perlas and Roukhomovsky mathematical models
  Interventions: Device: Gastric ultrasonography

INTERVENTIONS:
Device: Gastric ultrasonography — It seems like the text you provided is already in Turkish and it appears to be written in an academic style. If you want this text to be translated to English in an academic language, it would be:
  Ultrasonographic evaluation of gastric contents in Diabetic and Non-Diabetic term pregnancies

SUMMARY:
Perioperative aspiration is particularly concerning in pregnant women due to anatomical changes. To mitigate this risk, pre-anesthetic fasting is recommended, with varying guidelines. Gastric ultrasound can non-invasively assess stomach contents, and mathematical models help estimate stomach volumes using the gastric antral cross-sectional area (CSA).

This study aims to compare CSA and estimated gastric volumes through ultrasound in fasting diabetic and non-diabetic pregnant women scheduled for cesarean section, as diabetes may affect stomach fullness. Additionally, it will investigate the relation between demographic and clinical variables and CSA values.

This research can shed light on diabetes' influence on aspiration risk in pregnancy and evaluate fasting guidelines, underscoring the significance of gastric ultrasound.

DETAILED DESCRIPTION:
Perioperative aspiration of stomach contents is rare but is a serious complication of anesthesia and is associated with high morbidity and mortality. In pregnant women, it is known that the risk of aspiration is high even after standard preoperative fasting, due to anatomical changes such as the displacement of the stomach by pressure from the uterus, the sliding of the lower segment of the esophagus into the thorax, the relaxation of the lower esophageal sphincter, and the smooth muscle relaxation induced by progesterone.

In cases where regional anesthesia is contraindicated, various measures, including prokinetic and antacid medications, rapid-sequence anesthetic induction, and tracheal intubation, are used to reduce the risk and severity of pulmonary aspiration. However, the most commonly used measure is pre-anesthetic fasting in the patient. The European Society of Anaesthesiology (ESA) recommends fasting for ≥2 hours after clear liquids and 6 hours after light meals before elective surgery, including in pregnant patients.

The American Society of Anesthesiologists (ASA), on the other hand, recommends longer fasting times in pregnant patients without specifying the duration.

Aspiration risk in pregnant women is multifactorial. The type and volume of stomach contents, which are the main risk factors for aspiration, can be easily evaluated preoperatively with gastric ultrasonography. The presence of solids or thick liquids indicates a high risk of aspiration, independent of stomach volume.

However, in the presence of clear liquid, the risk of aspiration is generally linked to the volume of liquid in the stomach. The clear stomach volume limits that increase the risk of aspiration are controversial.

Some studies have shown that fasted patients generally have a gastric residual volume of up to 1.5 mL kg-1, and this value is used to determine the stomach at high risk for aspiration.

Gastric ultrasound assessment is an easy method that can be applied non-invasively at the bedside for evaluating gastric contents before anesthesia induction in the obstetric population. By measuring the gastric antral cross-sectional area (CSA), it may be possible to identify patients at risk for pulmonary aspiration with an estimate of stomach volume. Studies have shown the presence of a good linear correlation between antral CSA and stomach volume, not only in non-pregnant individuals but also in pregnant individuals.

Additionally, antral CSA measurement can indirectly differentiate small gastric volumes, consistent with initial gastric secretions, ≤1.5 mL kg-1, from larger volumes that may be associated with increased pulmonary aspiration risk.

Perlas et al. have developed a simple mathematical model based on the patient's age and antral CSA value measured in the right lateral position to calculate the volume of stomach fluid in non-pregnant adults and children.

Recently, two different mathematical models have been defined by Arzola et al.and Roukhomovsky et al. to estimate stomach volumes in pregnant patients. In this study, the investigators will use the mathematical formula developed by Roukhomovsky et al., as this model evaluates the presence of any stomach content, liquid or solid, rather than the volume of fluid swallowed as standard, with MR. Additionally, the model of Perlas et al., which is widely used in clinical practice and has been verified by studies, will be used.

It is accepted that there is gastroparesis in 9.9% - 76% of diabetic patients. Garg et al. in their prospective case-control study including 103 non-pregnant patients found that diabetic patients had higher gastric antral CSA and gastric volumes than non-diabetic patients. Sharma et al. have also shown that fasting for more than 6-10 hours does not guarantee an empty stomach and patients with comorbid diseases such as diabetes mellitus (DM), obesity are prone to having risky stomach contents. In DM patients, a significant increase in CSA in both supine and right lateral decubitus positions was detected compared to non-DM patients. Additionally, in the same study, it was found that as BMI increased from 25 to 35, there was a steady increase in CSA in both supine and right lateral decubitus positions. However, these studies were conducted in non-pregnant patients and the investigators did not come across similar studies conducted with diabetic pregnant women in the literature.

Recently, gastric ultrasound scanning before anesthesia in cases where the fasting state is unclear or unknown in the pregnant patient population, which is known to be more risky in terms of pulmonary aspiration, is recommended although not yet widespread in practical use. The effect of diabetes on stomach fullness is still controversial. There are many studies on gastric ultrasound evaluation in pregnant women, but the investigators have not come across a study comparing diabetic pregnant women with non-diabetics. This study was planned based on the idea that the presence of diabetes in pregnant women could further increase the risk of pulmonary aspiration. The primary aim of this research is to compare the antral cross-sectional area (CSA) with gastric ultrasound and estimated gastric volumes calculated with 2 mathematical models in fasting diabetic and non-diabetic term pregnant women who will be taken for cesarean section.

The secondary aim is to determine the relationship between demographic and clinical variables and gastric antral CSA values in fasting term pregnant women. the investigators believe that our study will contribute to the literature with its originality and results. Additionally, the investigators believe that our study will provide insight into the effectiveness of fasting guidelines in these patient groups and the necessity of gastric ultrasound scanning."

ELIGIBILITY:
Inclusion Criteria:

* Patients belonging to American Society of Anesthesiology (ASA) physical status class II-III.
* Aged between 18 and 40 years.
* Gestational age greater than 37 weeks.
* BMI< 35 kg/m2

Exclusion Criteria:

* Patients belonging to American Society of Anesthesiology (ASA) physical status class III-IV.
* Patients under the age of 18.
* Patients taken to surgery on an emergency basis.
* Relatives of patients who do not provide consent.
* Pregnant patients with upper gastrointestinal (GI) diseases and pathologies.
* Body Mass Index (BMI) greater than 35 kg/m2.
* Patients with a history of using medications that affect gastrointestinal motility (e.g., opioids).
* Severe organ dysfunction.
* Pre-existing neurological deficits.
* Intellectual disabilities.
* Anatomical deformities.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Term pregnant women
Study Population: It is planned to include 80 diabetic and non-diabetic patients aged 18-40 years, belonging to the ASA (American Society of Anesthesiologists) physical status class II-III, who are scheduled for elective cesarean surgery. Randomization will be carried out using a sealed envelope method. Two groups, each comprising 40 patients, will be formed and evaluated with preoperative gastric ultrasound.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-07-26 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
Antral cross-sectional area (in square centimeters) | 2 months
  Ultrasonographic gastric antral cross-sectional area in square centimeters=(D1 × D2 × π)/4. Anteroposterior diameter of the antrum from serosa to serosa: D1 (centimeters), craniocaudal diameter: D2 (centimeters)
Perlas equation for gastric volume (mL) | 2 months
  Perlas Gastric residual volume (mL) = 27.0 + 14.6 x right lateral CSA (cm2) - 1.28 x age (years).
Roukhomovsky equation for gastric volume (mL) | 2 month
  Roukhomovsky Gastric residual volume (mL) = 0.18 x right lateral CSA (mm2) + 0.11 x semi-recumbent CSA (mm2) - 62.4

SECONDARY OUTCOMES:
Relationship between demographic/clinical features and CSA (cm2) / Perlas GV (mL/kg) / Roukhomovsky GV (mL/kg) values. | 2 months
  The examination of the correlation/relationship between age (years), BMI (weight and height will be combined to report BMI in kg/m2), ASA (II-III), gestational age (weeks), fasting time for liquids (hour) and solids (hour), and supine CSA, right lateral CSA, Perlas GV (mL/kg) and Roukhomovsky GV (mL/kg) values.

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Kesici, Assoc. Prof., Principal Investigator — Sisli Etfal
Locations (1):
- Sisli Hamidiye Etfal Training and Research Hospital, Sarıyer, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] MENDELSON CL. The aspiration of stomach contents into the lungs during obstetric anesthesia. Am J Obstet Gynecol. 1946 Aug;52:191-205. doi: 10.1016/s0002-9378(16)39829-5. No abstract available. PMID 20993766
- [Result] Smith I, Kranke P, Murat I, Smith A, O'Sullivan G, Soreide E, Spies C, in't Veld B; European Society of Anaesthesiology. Perioperative fasting in adults and children: guidelines from the European Society of Anaesthesiology. Eur J Anaesthesiol. 2011 Aug;28(8):556-69. doi: 10.1097/EJA.0b013e3283495ba1. PMID 21712716
- [Result] Practice Guidelines for Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration: Application to Healthy Patients Undergoing Elective Procedures: An Updated Report by the American Society of Anesthesiologists Task Force on Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration. Anesthesiology. 2017 Mar;126(3):376-393. doi: 10.1097/ALN.0000000000001452. No abstract available. PMID 28045707
- [Result] El-Boghdadly K, Wojcikiewicz T, Perlas A. Perioperative point-of-care gastric ultrasound. BJA Educ. 2019 Jul;19(7):219-226. doi: 10.1016/j.bjae.2019.03.003. Epub 2019 Apr 24. No abstract available. PMID 33456894
- [Result] Van de Putte P, Perlas A. Ultrasound assessment of gastric content and volume. Br J Anaesth. 2014 Jul;113(1):12-22. doi: 10.1093/bja/aeu151. Epub 2014 Jun 3. PMID 24893784
- [Result] Van de Putte P, Vernieuwe L, Perlas A. Term pregnant patients have similar gastric volume to non-pregnant females: a single-centre cohort study. Br J Anaesth. 2019 Jan;122(1):79-85. doi: 10.1016/j.bja.2018.07.025. Epub 2018 Aug 29. PMID 30579409
- [Result] Arzola C, Perlas A, Siddiqui NT, Carvalho JCA. Bedside Gastric Ultrasonography in Term Pregnant Women Before Elective Cesarean Delivery: A Prospective Cohort Study. Anesth Analg. 2015 Sep;121(3):752-758. doi: 10.1213/ANE.0000000000000818. PMID 26097988
- [Result] Perlas A, Chan VW, Lupu CM, Mitsakakis N, Hanbidge A. Ultrasound assessment of gastric content and volume. Anesthesiology. 2009 Jul;111(1):82-9. doi: 10.1097/ALN.0b013e3181a97250. PMID 19512861
- [Result] Perlas A, Van de Putte P, Van Houwe P, Chan VW. I-AIM framework for point-of-care gastric ultrasound. Br J Anaesth. 2016 Jan;116(1):7-11. doi: 10.1093/bja/aev113. Epub 2015 May 7. No abstract available. PMID 25951832
- [Result] Perlas A, Mitsakakis N, Liu L, Cino M, Haldipur N, Davis L, Cubillos J, Chan V. Validation of a mathematical model for ultrasound assessment of gastric volume by gastroscopic examination. Anesth Analg. 2013 Feb;116(2):357-63. doi: 10.1213/ANE.0b013e318274fc19. Epub 2013 Jan 9. PMID 23302981
- [Result] Arzola C, Perlas A, Siddiqui NT, Downey K, Ye XY, Carvalho JCA. Gastric ultrasound in the third trimester of pregnancy: a randomised controlled trial to develop a predictive model of volume assessment. Anaesthesia. 2018 Mar;73(3):295-303. doi: 10.1111/anae.14131. Epub 2017 Dec 19. PMID 29265187
- [Result] Roukhomovsky M, Zieleskiewicz L, Diaz A, Guibaud L, Chaumoitre K, Desgranges FP, Leone M, Chassard D, Bouvet L; AzuRea, CAR'Echo Collaborative Networks. Ultrasound examination of the antrum to predict gastric content volume in the third trimester of pregnancy as assessed by MRI: A prospective cohort study. Eur J Anaesthesiol. 2018 May;35(5):379-389. doi: 10.1097/EJA.0000000000000749. PMID 29210844
- [Result] Jellish WS, Kartha V, Fluder E, Slogoff S. Effect of metoclopramide on gastric fluid volumes in diabetic patients who have fasted before elective surgery. Anesthesiology. 2005 May;102(5):904-9. doi: 10.1097/00000542-200505000-00007. PMID 15851875
- [Result] Garg H, Podder S, Bala I, Gulati A. Comparison of fasting gastric volume using ultrasound in diabetic and non-diabetic patients in elective surgery: An observational study. Indian J Anaesth. 2020 May;64(5):391-396. doi: 10.4103/ija.IJA_796_19. Epub 2020 May 1. PMID 32724247
- [Result] Sharma G, Jacob R, Mahankali S, Ravindra MN. Preoperative assessment of gastric contents and volume using bedside ultrasound in adult patients: A prospective, observational, correlation study. Indian J Anaesth. 2018 Oct;62(10):753-758. doi: 10.4103/ija.IJA_147_18. PMID 30443057